CLINICAL TRIAL: NCT00000690
Title: Single Dose Pharmacokinetics of Oral Dextran Sulfate (UA001) and Intravenous Dextran Sulfate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 078; 11053 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Reference Values; Infusions, Intravenous; Intestinal Absorption; Dextran Sulfate; Administration, Oral; Blood Coagulation
MeSH Terms: conditions — HIV Infections; Thrombosis | interventions — Dextran Sulfate

INTERVENTIONS:
Drug: Dextran sulfate

SUMMARY:
To evaluate how the drug dextran sulfate (DS) is absorbed by the stomach and intestines when taken by mouth. To evaluate its effect on blood coagulation.

DS has been reported to have anti-HIV activity. However, it is not known how much of the drug is absorbed into the bloodstream and can be used by the body when DS is taken by mouth.

DETAILED DESCRIPTION:
DS has been reported to have anti-HIV activity. However, it is not known how much of the drug is absorbed into the bloodstream and can be used by the body when DS is taken by mouth.

On 2nd day of hospitalization, each volunteer receives an oral dose of DS. Over the next 24 hours, 15 blood samples are obtained (from 15 separate needle sticks). On 4th day, each volunteer is given an injection of DS into vein. 18 blood samples are obtained. Blood is withdrawn before the infusion, at the end of the infusion, and 30 and 60 minutes after the infusion. All urine is collected.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Volunteers with any of the following are excluded:

* Disorders of coagulation or disorders of plasma lipids.
* Allergy to dextran sulfate, other sulfates, other dextrans.

Concurrent Medication:

Excluded:

* Volunteers who anticipate need for medication during study.

Volunteers with any of the following are excluded:

* Disorders of coagulation or disorders of plasma lipids.
* Allergy to dextran sulfate, other sulfates, other dextrans.

Prior Medication:

Excluded within 2 weeks of study entry:

* Any medication.

Risk Behavior:

Excluded:

* Ingestion of alcohol within 48 hours prior to study.
* History of recent drug or alcohol abuse.
* Disorders of coagulation or disorders of plasma lipids.
* Allergy to dextran sulfate, other sulfates, other dextrans.

Volunteers selected are:

* In good general health as determined by screening history, physical examination, and laboratory panel within established limits of normal for hospital laboratory.
* Consenting volunteers.
* Available for 6 days of continuous hospitalization.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6
Dates: Study Completion 1989-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P Lietman, Study Chair; KJ Lorentsen, Study Chair; CW Hendrix, Study Chair; JM Collins, Study Chair; DM Kornhauser, Study Chair; BG Petty, Study Chair
Locations (1):
- Johns Hopkins Hosp, Baltimore, Maryland, United States

REFERENCES:
- [Background] Flexner C, Barditch-Crovo PA, Kornhauser DM, Farzadegan H, Nerhood LJ, Chaisson RE, Bell KM, Lorentsen KJ, Hendrix CW, Petty BG, et al. Pharmacokinetics, toxicity, and activity of intravenous dextran sulfate in human immunodeficiency virus infection. Antimicrob Agents Chemother. 1991 Dec;35(12):2544-50. doi: 10.1128/AAC.35.12.2544. PMID 1810188
- [Background] Hiebert LM, Wice SM, Jaques LB, Williams KE, Conly JM. Orally administered dextran sulfate is absorbed in HIV-positive individuals. J Lab Clin Med. 1999 Feb;133(2):161-70. doi: 10.1016/s0022-2143(99)90009-4. PMID 9989768
- [Background] Lorentsen KJ, Hendrix CW, Collins JM, Kornhauser DM, Petty BG, Klecker RW, Flexner C, Eckel RH, Lietman PS. Dextran sulfate is poorly absorbed after oral administration. Ann Intern Med. 1989 Oct 1;111(7):561-6. doi: 10.7326/0003-4819-111-7-561. PMID 2476054